CLINICAL TRIAL: NCT02252055
Title: A Phase I/II Monocentric Trial of Cellular Immunotherapy Based on Autologous Tolerogenic Dendritic Cells (ATDCs) Administration in Patients With Renal Insufficiency Receiving as First Transplantation a Kidney Transplant From a Living-donor.
Brief Title: The ONE Study ATDC Trial
Acronym: ONEatDC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC13_0441
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Renal Failure, End Stage
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ATDC Treatment (Experimental): ATDC treatment (1 x 106 cells/kg BW slow peripheral venous) occurs the day before transplantation.
  Recipients also receive prednisolone, Mycophenolate Mofetil and tacrolimus, as detailed below :
  Prednidolone :
  * D 0: 500 mg IV
  * D 1: 125 mg IV
  * D 2 to 14: 20.0 mg/d
  * Wk 3 to 4: 15.0 mg/d
  * Wk 5 to 8: 10.0 mg/d
  * Wk 9 to 12: 5.0 mg/d
  * Wk 13 to 14: 2.5 mg/d
  * Wk 15 to End:Cessation
  MMF (or biologic equiv.):
  * D -7 to -2: 500 mg/d (250mg 2x/d)
  * D -1 to 14: 2000 mg/d
  * Wk 3 to 36: 1000 mg/d
  * Wk 37 to 40: 750 mg/d
  * Wk 41 to 44: 500 mg/d
  * Wk 45 to 48: 250 mg/d
  * Wk 49 to End:Cessation Note : MMF tapering will only happen if the 36-week protocol biopsy shows no signs of subclinical rejection and there is evidence of declining renal function or if the clinician has any other concern about MMF dose reduction.
  Tacrolimus :
  * ≤ 48 h pre-Tx to D 14: 3-12 ng/ml
  * Wk 3 to 12: 3-10 ng/ml
  * Wk 13 to 36: 3-8 ng/ml
  * Wk 37 to End: 3-6 ng/ml
  Interventions: Biological: ATDC_Nantes

INTERVENTIONS:
Biological: ATDC_Nantes — ATDC treatment (1 x 106 cells/kg BW slow peripheral venous) occurs the day before transplantation into recipients also recipients of a living donor renal transplantation.
  Recipients also receive prednisolone, Mycophenolate Mofetil and tacrolimus background immunosuppression ( as described in detail in the arm description)

SUMMARY:
To collect evidence of the safety of administering autologous tolerogenic dendritic cells (ATDC) preparations to living-donor renal transplant recipients in the context of an international European Union funded consortium aimed at evaluationg cellular immunotherapy in solid organ transplantation (The ONE Study). It is anticipated that immune regulation induced by ATDC therapy can evntually be used to reduce the need for conventional immunosuppression in transplant recipients.

DETAILED DESCRIPTION:
Decades of immunosuppressive drug development have produced an array of powerful pharmacological agents, but the various drawbacks associated with these treatments leaves considerable room for improvement. By harnessing the power of suppressive mechanisms in the human immune system, regulatory cell therapy may be able to support peripheral tolerance and induce a level of donor-specific unresponsiveness that allows for a reduction in the use of conventional immunosuppression in organ transplant recipients. Several alternative regulatory cell types have been identified as potential adjunct immunotherapies for solid organ transplantation and are now approaching a stage of development that would allow clinical testing in an early-stage trial. The ONE Study aims to answer the question as whether ATDC treatment, or immunoregulatory cell-based therapy in general, has any place in the clinical management of solid organ transplant recipients.

ELIGIBILITY:
RECIPIENT

Inclusion Criteria:

1. Chronic renal insufficiency necessitating kidney transplantation and approved to receive a primary kidney allograft from a living donor
2. Aged at least 18 years
3. Able to commence the immunosuppressive regimen at the protocol-specified time point
4. Willing and able to participate in The ONE Study IM and HEC subprojects
5. Eligible for leucapheresis prior to organ transplantation
6. Signed and dated written informed consent

Exclusion Criteria:

1. Patient has previously received any tissue or organ transplant other than the planned kidney graft
2. Known contraindication to the protocol-specified treatments / medications (like known allergies to heparin)
3. Genetically identical to the prospective organ donor at the HLA loci (A.B.DR 0 mismatch)
4. PRA grade > 0 within 6 months prior to enrolment
5. Previous treatment with any desensitisation procedure (with or without IVIg)
6. Concomitant malignancy or history of malignancy within 5 years prior to planned study entry (excluding successfully-treated non-metastatic basal/squamous cell carcinoma of the skin)
7. ABO incompatibility
8. Presence of DSA (donor specific antibodies) detected by luminex prior transplantation
9. Evidence of significant local or systemic infection
10. HIV-positive, EBV-negative or suffering chronic viral hepatitis, syphilis serology- positive
11. Significant liver disease, defined as persistently elevated AST and/or ALT levels > 2 x ULN (Upper Limit of Normal range)
12. Malignant or pre-malignant haematological conditions
13. Any uncontrolled medical condition or concurrent disease that could interfere with the study objectives
14. Any condition which, in the judgement of the Investigator, would place the subject at undue risk
15. Ongoing treatment with systemic immunosuppressive drugs at inclusion (despite corticoids lower than 10 mg)
16. Participation in another clinical trial during the study or within 28 days prior to planned study entry
17. Exposure to an investigational product during the study or within 28 days prior to planned study entry
18. Female patients of child-bearing potential with a positive pregnancy test at enrolment and F01
19. Female patients who are breast-feeding
20. All female patients of child-bearing potential* UNLESS:

    1. The patient is willing to maintain a highly effective method of birth control** for the duration of the study
    2. The career, lifestyle, or sexual orientation of the patient ensures that there is no risk of pregnancy for the duration of the study (at the discretion of the Investigator)
21. Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up visit schedule
22. Any form of substance abuse, psychiatric disorder, or other condition that, in the opinion of the Investigator, may invalidate communication with the Investigator and/or designated study personnel
23. Patients unable to freely give their informed consent (e.g. individuals under legal guardianship).

    Criteria specific to the infusion of the ATDC_Nantes:
24. Any pro-coagulant disposition, as evidenced by a past history of thromboembolic disease or abnormal laboratory coagulation parameters which, in the judgement of the Investigator, would place the subject at undue risk
25. Any condition resulting in a substantial reduction in the volume of the pulmonary vasculature or an increase in the pulmonary vascular resistance. Any disease or disease process leading to substantially elevated pulmonary arterial pressure (as evidenced by electrocardiography, echocardiography, radiology or cardiac catheterisation) or right heart hypertrophy or dysfunction
26. Known atrial or ventricular septal defects posing a risk of paradoxical embolism of infused cells or cell aggregates
27. Known hypersensitivity to any component of the cell product or components used in the manufacture of the cell product.

DONOR

Inclusion Criteria:

1. Eligible for live kidney donation
2. Willing and able to provide a blood sample for The ONE Study IM Subproject
3. Willing to provide personal and medical/biological data for the trial analysis
4. Signed and dated written informed consent

Exclusion Criteria:

1. Genetically identical to the prospective organ recipient at the HLA loci (A.B.DR 0 mismatch)
2. Exposure to any investigational agents at the time of kidney donation, or within 28 days prior to kidney donation
3. Any form of substance abuse, psychiatric disorder, or other condition that, in the opinion of the Investigator, may invalidate communication with the Investigator and/or designated study personnel
4. Subjects unable to freely give their informed consent (e.g. individuals under legal guardianship).
5. ABO incompatibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-03-19 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
Incidence of biopsy-confirmed acute rejection (BCAR) | 60 weeks

SECONDARY OUTCOMES:
Time to first acute rejection episode | 60 weeks
Severity of acute rejection episodes | 60 weeks
  based on response to treatment and histological scoring
Total immunosuppressive burden | 60 weeks
  assessed at last study visit
Incidence of patients treated for subclinical acute rejection on the basis of histopathological findings | 60 weeks
Prevention of chronic graft dysfunction (chronic rejection or IF/TA) | 60 weeks
  assessed by clinical (impairment of GFR) and histopathological (Banff staging) measures.
Incidence of post-transplant dialysis, inclusion on the transplant waiting list or re-transplantation following graft loss through rejection (acute or chronic). | 60 weeks
Avoidance of drug-related complications by immunosuppressant reduction | 60 weeks
Incidence of embolic pulmonary complications and other embolic events | 60 weeks
Incidence of immunological reactions resulting in anaphylactoid reactions, immediate cardiovascular compromise or other acute organ failure | 1 week
Biochemical disturbances caused by cell infusion | 1 week
Over-suppression of the immune system assessed by the incidence of major and/or opportunistic infections, especially CMV, EBV and polyoma virus | 1 week
Over-suppression of the immune system assessed by the incidence of neoplasia. | 1 week
Immunological condition of study patients w | 60 weeks
  an extensive immune monitoring program has been established in the ONE Study

OTHER OUTCOMES:
Incidence of malignancies arising directly from ATDC_Nantes | 60 weeks
ii) incidence of autoimmune disorders | 60 weeks
Incidence of inflammatory pathologies | 60 weeks
Incidence of anaemia, cytopaenia or biochemical disturbances unrelated to the function of the transplanted kidney. | 60 weeks
A Health-Economic Subproject will evaluate the health-related quality-of-life of trial patients using patient-reported outcome measures. | 60weeks
  This subproject will also calculate the cost-effectiveness of ATDC_Nantes to review the financial implications of cellular immunotherapy as a practical and routine clinical prescription.

CONTACTS AND LOCATIONS:
Overall Officials: Edward K Geissler, PhD, Study Director — University Hospital Regensburg
Locations (1):
- Nantes University hospital, Nantes, France

REFERENCES:
- [Background] Geissler EK. The ONE Study compares cell therapy products in organ transplantation: introduction to a review series on suppressive monocyte-derived cells. Transplant Res. 2012 Sep 28;1(1):11. doi: 10.1186/2047-1440-1-11. No abstract available. PMID 23369457
- [Derived] Moreau A, Kervella D, Bouchet-Delbos L, Braudeau C, Saiagh S, Guerif P, Limou S, Moreau A, Bercegeay S, Streitz M, Sawitzki B, James B, Harden PN, Game D, Tang Q, Markmann JF, Roberts ISD, Geissler EK, Dreno B, Josien R, Cuturi MC, Blancho G; DIVAT consortium. A Phase I/IIa study of autologous tolerogenic dendritic cells immunotherapy in kidney transplant recipients. Kidney Int. 2023 Mar;103(3):627-637. doi: 10.1016/j.kint.2022.08.037. Epub 2022 Oct 26. PMID 36306921
- [Derived] Sawitzki B, Harden PN, Reinke P, Moreau A, Hutchinson JA, Game DS, Tang Q, Guinan EC, Battaglia M, Burlingham WJ, Roberts ISD, Streitz M, Josien R, Boger CA, Scotta C, Markmann JF, Hester JL, Juerchott K, Braudeau C, James B, Contreras-Ruiz L, van der Net JB, Bergler T, Caldara R, Petchey W, Edinger M, Dupas N, Kapinsky M, Mutzbauer I, Otto NM, Ollinger R, Hernandez-Fuentes MP, Issa F, Ahrens N, Meyenberg C, Karitzky S, Kunzendorf U, Knechtle SJ, Grinyo J, Morris PJ, Brent L, Bushell A, Turka LA, Bluestone JA, Lechler RI, Schlitt HJ, Cuturi MC, Schlickeiser S, Friend PJ, Miloud T, Scheffold A, Secchi A, Crisalli K, Kang SM, Hilton R, Banas B, Blancho G, Volk HD, Lombardi G, Wood KJ, Geissler EK. Regulatory cell therapy in kidney transplantation (The ONE Study): a harmonised design and analysis of seven non-randomised, single-arm, phase 1/2A trials. Lancet. 2020 May 23;395(10237):1627-1639. doi: 10.1016/S0140-6736(20)30167-7. PMID 32446407
- See also: Related Info — http://www.onestudy.org